CLINICAL TRIAL: NCT06360406
Title: Real-World Treatment Study of Koselugo (Selumetinib)
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1346R00009
Record Dates: First submitted 2024-04-08; First posted 2024-04-11 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Neurofibromatosis 1; Neurofibroma, Plexiform
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibroma, Plexiform

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
As part of a post-approval commitment, the Korean health authority requests a study to characterize safety and effectiveness in patients treated with Koselugo (Selumetinib), an oral selective inhibitor of MAPK kinase (MEK) 1 and 2, by physicians in routine clinical practice settings. This study is designed to assess the known safety profile or identify previously unsuspected adverse reactions and evaluate the effectiveness of Koselugo under conditions of routine daily medical practice in Korea.

This study will provide information on the Korean patient population that is treated with the study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Patients treated with Koselugo (Selumetinib) under the approved label in South Korea
2. Provision of signed and dated written informed consent by the patient or legally acceptable representative

Exclusion Criteria:

1. Patients treated with Koselugo (Selumetinib) under the approved label in South Korea
2. Provision of signed and dated written informed consent by the patient or legally acceptable representative

Ages: 3 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with Koselugo (Selumetinib) under the approved label in South Korea.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-06-15 (Actual); Primary Completion 2031-09-30 (Estimated); Study Completion 2031-09-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) rate | 1 year
  To assess the safety (Adverse events (AEs), serious AEs (SAEs), adverse drug reactions (ADRs), serious ADRs (SADRs), unexpected AEs/ADRs) of the study drug for patients prescribed with the study drug under the approved indication(s) in Korea
Physeal dysplasia occurance rate | 1 year
  To assess the safety of the study drug for patients prescribed with the study drug under the approved indication(s) in Korea

SECONDARY OUTCOMES:
Descriptive analysis with the physician qualitative assessments by overall disease status of NF-1 and status of clinically significant PNs, respectively. - Improving - Progression - Stable | 1 year
  To assess the effectiveness of the study drug for patients prescribed with the study drug under the approved indication(s) in Korea

CONTACTS AND LOCATIONS:
Locations (9):
- South Korea (9):
  - Research Site, Busan
  - Research Site, Chungcheongbuk-do
  - Research Site, Daejeon
  - Research Site, Gyeonggi-do
  - Research Site, Incheon
  - Research Site, Jeonnam
  - Research Site, Seoul
  - Research Site, Wŏnju
  - Research Site, Yangsan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/